CLINICAL TRIAL: NCT05194839
Title: A Randomized, Double-blind, Placebo-controlled, Dose Ranging Phase 2 Study to Evaluate the Efficacy and Safety of RIST4721 in Subjects With Palmoplantar Pustulosis
Brief Title: A Phase 2b Study to Evaluate RIST4721 in Palmoplantar Pustulosis (PPP)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to safety findings in ongoing Phase 2 trials.
Sponsor: Aristea Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIST4721-202
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Palmoplantar Pustulosis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RIST4721 400 mg (Experimental): RIST4721 400 mg: 4 active (100 mg) tablets once daily for 12 weeks
  Interventions: Drug: RIST4721
- RIST4721 200 mg (Experimental): RIST4721 200 mg: 2 active (100 mg) tablets + 2 placebo tablets once daily for 12 weeks
  Interventions: Drug: RIST4721; Drug: Placebo
- Placebo (Placebo Comparator): Placebo: 4 placebo tablets once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RIST4721 — RIST4721 tablets, 100 mg are blue, oval, biconvex film-coated tablets
  Arms: RIST4721 200 mg; RIST4721 400 mg
Drug: Placebo — Matching placebo
  Arms: Placebo; RIST4721 200 mg

SUMMARY:
A 12-week Randomized, Double-blind, Placebo-controlled, Dose Ranging Phase 2 Study to Evaluate the Efficacy and Safety of RIST4721 in Subjects with Palmoplantar Pustulosis followed by an Open-label Extension Phase.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months history of moderate or severe PPP, as defined by PPPASI ≥12 and PPPGA ≥3 at screening
* Males and females must be willing to use birth control as indicated

Exclusion Criteria:

* Moderate to severe psoriasis covering ≥10% of total body surface area (BSA) at screening
* Breastfeeding or pregnant
* Known immunodeficiency or subject is immunocompromised
* Active/latent infection with HBV, HCV, HIV, SARS-CoV-2 or TB
* Any topical medications for PPP excluding emollients within two weeks of randomization and systemic therapies (including phototherapy) within 4 weeks of randomization

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (19):
  - Total Skin & Beauty Dermatology Center, PC, Birmingham, Alabama
  - Dermatology Trial Associates, Bryant, Arkansas
  - Cosmetic Laser Dermatology, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Driven Research LLC, Coral Gables, Florida
  - Encore Medical Research, LLC, Hollywood, Florida
  - Tory Sullivan, MD PA, North Miami Beach, Florida
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DS Research, Louisville, Kentucky
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Washington University School of Medicine-Dermatology, St Louis, Missouri
  - Skin Specialists, PC (Schlessinger MD), Omaha, Nebraska
  - ALLCUTIS Research, LLC., Portsmouth, New Hampshire
  - Aventiv Research Inc., Dublin, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
- Canada (6):
  - Alberta DermaSurgery Centre, Edmonton, Alberta
  - Vida Dermatology, Edmonton, Alberta
  - Central Alberta Research Clinic (CARe Clinic), Red Deer, Alberta
  - SimcoDerm Medical and Surgical, Barrie, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Centre De Recherche Dermatologique Du Quebec Metropolitan Inc., Québec
- Czechia (3):
  - Kožní ambulance Kutná Hora, s.r.o., Kutná Hora
  - Clintrial s.r.o, Prague
  - Praglandia s.r.o., Prague
- Germany (11):
  - Universitätsklinikum Augsburg Klinik für Dermatologie und Allergologie, Augsburg
  - Fachklinik Bad Bentheim Fachbereich Dermatologie und Allergologie, Bad Bentheim
  - Uniklinikum Dresden Klinik und Poliklinik für Dermatologie, Dresden
  - Universitätsklinikum Erlangen Hautklinik, Erlangen
  - TFS Trial Form Support GmbH SCIderm - Zentrum für klinische Studien, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel [Zentrum für entzundliche Hauterkrankungen] Klinik für Dermatologie, Venerologie und Allergologie, Kiel
  - Hautarztpraxis Mahlow, Mahlow
  - Klinikum der Universität München Klinik und Poliklinik der Dermatologie und Allergologie Der Universität München, München
  - Universitaetsklinikum Muenster, Münster
  - KliFOs - Klinische Forschung Osnabrück, Osnabrück
  - Hautarztpraxis Dres. Leitz & Kollegen, Stuttgart
- Hungary (4):
  - Semmelweis University, Department of Dermatology, Venerology and Dermatooncology, Budapest
  - University of Debrecen, Dermatology Department, Debrecen
  - Bács-Kiskun Megyei KórházSzegedi Tudományegyetem Általános Orvostudományi Kar Oktató Kórháza Bórgyógyászati Szakrendelés, Kecskemét
  - University of Pecs, Department of Dermatology, Venerology and Oncodermatology, Pécs
- Poland (7):
  - Diamond Clinic Spolka z ograniczona odpowiedzialnoscia, Krakow
  - Clinical Best Solutions, Lublin
  - Luxderm Specjalistyczny Gabinet Dermatologiczny, Lublin
  - Luxderm Specjalistyczny Gabinet Dermatologiczny, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Przychodnia Lekarsko-Psychologinczna Matusiak Spółka Partnerska, Wroclaw
  - DermMedica Sp. z o.o., Wroclaw
- Salford Care Organisation, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RIST4721 400 mg | RIST4721 200 mg | Placebo
Started | 27 | 26 | 26
Completed | 12 | 13 | 12
Not Completed | 15 | 13 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RIST4721 400 mg | RIST4721 200 mg | Placebo | Total
Number analyzed (Participants) | 27 | 26 | 26 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 22 | 20 | 63
  >=65 years | 6 | 4 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 19 | 65
  Male | 4 | 3 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 26 | 26 | 25 | 77
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving a 50% Reduction in PPPASI Score
Description: In the Palmoplantar Pustulosis Psoriasis Area and Severity Index (PPPASI), the left palm, right palm, left foot, and right foot are assessed based on 3 target symptoms: erythema, desquamation (scaling), and pustules, as seen on the day of the examination. The severity of each sign is assessed using a 5-point scale (0 = not present, 1 = slight, 3 = moderate, 4 = severe, 5 = very severe). The affected area within a given anatomic site (left palm, right palm, left foot, and right foot) is estimated as a percentage of the total area of that anatomic site and assigned a numerical value according to the degree of PPP involvement (0 = no involvement, 2 = 10 to less than 30% involvement, 3 = 30 to less than 50% involvement, 4 = 50 to less than 70% involvement, 5 = 70 to less than 90% involvement, 6 = 90 to less than 100% involvement). PPPASI score for palms and soles is obtained using a formula and can vary from 0 (absence of disease) to 72 (most severe disease).
Time Frame: Baseline to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | RIST4721 400 mg | RIST4721 200 mg | Placebo
Number analyzed (Participants) | 12 | 13 | 12
Participants | 6 | 3 | 5

2. Secondary Outcome: Absolute Change From Baseline in PPPGA
Time Frame: Baseline to Week 12
Reporting Status: Not Posted

3. Secondary Outcome: Absolute Change From Baseline in PPPASI
Time Frame: Baseline to Week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through end of Week 12 (blinded treatment) and up to 4 weeks of follow-up.
Arm/Group | RIST4721 400 mg | RIST4721 200 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/26 | 0/26
Other Adverse Events (participants affected / at risk) | 18/27 | 17/26 | 18/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIST4721 400 mg (N=27) | RIST4721 200 mg (N=26) | Placebo (N=26)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RIST4721 400 mg (N=27) | RIST4721 200 mg (N=26) | Placebo (N=26)
Nasopharyngitis (Infections and infestations) | 1 | 3 | 4
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 1
Covid-19 (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0
C-reactive protein increased (Investigations) | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 1 | 1
Urine odor abnormal (Renal and urinary disorders) | 1 | 3 | 0
Hypertension (Vascular disorders) | 2 | 0 | 1
Asymptomatic COVID-19 (Infections and infestations) | 1 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cystitis bacterial (Infections and infestations) | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Viral diarrhoea (Infections and infestations) | 0 | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Invertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1
Vertigo (Nervous system disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 2 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT05194839/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT05194839/SAP_001.pdf